CLINICAL TRIAL: NCT00947115
Title: Follow-up Study to Evaluate the Long-term Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV (580299) Vaccine in Healthy Female Subjects
Brief Title: Evaluation of Long-term Immunogenicity and Safety of a Human Papillomavirus (HPV) Vaccine in Healthy Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112772; 2009-011357-41 (EudraCT Number)
Record Dates: First submitted 2009-07-16; First posted 2009-07-27 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Infections, Papillomavirus
Keywords: Cervical cancer; HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Blood Specimen Collection; Chorionic Villi Sampling

ARMS (3):
- Cervarix 15-25 years group (Experimental): Women, aged 15 to 25 at the time of primary vaccination, who were vaccinated with Cervarix intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule in the primary study HPV-014 (NCT00196937).
  Interventions: Procedure: Blood sampling; Procedure: Cervico-vaginal secretion (CVS) samples
- Cervarix 26-45 years group (Experimental): Women, aged 26 to 45 at the time of primary vaccination, who were vaccinated with Cervarix intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule in the primary study HPV-014 (NCT00196937).
  Interventions: Procedure: Blood sampling; Procedure: Cervico-vaginal secretion (CVS) samples
- Cervarix 46-55 years group (Experimental): Women, aged 46 to 55 at the time of primary vaccination, who were vaccinated with Cervarix intramuscularly into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule in the primary study HPV-014 (NCT00196937).
  Interventions: Procedure: Blood sampling; Procedure: Cervico-vaginal secretion (CVS) samples

INTERVENTIONS:
Procedure: Blood sampling — Blood samples were collected at Years 5, 6, 7, 8, 9 and 10.
Procedure: Cervico-vaginal secretion (CVS) samples — CVS samples were collected at Years 5, 6, 7, 8, 9 and 10 in subjects who volunteered for this procedure.

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the necessary cause of cervical cancer. This study is designed to evaluate the long-term immunogenicity and safety of the GSK Biologicals' 580299 HPV vaccine up to 10 years after administration of the first dose of HPV vaccine (Month 0) in primary study NCT00196937. This protocol posting deals with objectives & outcome measures of the extension phase from Year 5 to Year 10. The objectives & outcome measures of the primary phase and extension phase up to year 4 are presented in a separate protocol posting (NCT00196937).

DETAILED DESCRIPTION:
Subjects were aged 15-55 years at the time of entry into the primary study (NCT00196937). No vaccine was administered in this extension study.

Results on outcome measures describing analyses on other studies are not reported in this record. Please refer to the records mentioned in the respective outcome measure titles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believed that they could and would comply with the requirements of the protocol.
* A female who had been enrolled in NCT00196937 study and received three doses of HPV-16/18 vaccine.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) or planned use during the study period.
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs occurring less than three months prior to blood sampling.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Administration of immunoglobulins and/or any blood products within the three months preceding blood sampling.
* Administration or planned administration of any HPV vaccine, other than the three doses of HPV-16/18 vaccine administered in NCT00196937 study.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2015-02-03 (Actual); Study Completion 2015-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Berlin
- Poland (2):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Poznan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4512

REFERENCES:
- [Background] Schwarz T, Spaczynski M, Kaufmann A, Wysocki J, Galaj A, Schulze K, Suryakiran P, Thomas F, Descamps D. Persistence of immune responses to the HPV-16/18 AS04-adjuvanted vaccine in women aged 15-55 years and first-time modelling of antibody responses in mature women: results from an open-label 6-year follow-up study. BJOG. 2015 Jan;122(1):107-18. doi: 10.1111/1471-0528.13070. Epub 2014 Sep 11. PMID 25208608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at six centers in Germany and Poland.
Pre-assignment Details: Out of the 525 enrolled subjects, 1 subject was excluded for not receiving vaccination and the actual starting number was 524.
Period: Overall Study
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Started | 159 | 194 | 171
Completed | 142 | 172 | 156
Not Completed | 17 | 22 | 15
Not completed — Missed reporting interval | 3 | 4 | 2
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Migrated from study area | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Lost to Follow-up | 11 | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group | Total
Number analyzed (Participants) | 159 | 194 | 171 | 524
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data for Year 5 - Year 10
  Years | 25.7 (2.82) | 41.0 (6.02) | 54.4 (3.15) | 40.9 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants] — Data for Year 5 - Year 10
  Participants
    Female | 159 | 194 | 171 | 524
    Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data for Year 5 - Year 10
  Participants
    Black | 0 | 1 | 0 | 1
    White/Caucasian | 159 | 193 | 171 | 523

OUTCOME MEASURES:

1. Primary Outcome: Anti-Human Papillomavirus (Anti-HPV)-16/18 Antibody Titers in Serum at Years 5, 6 and 7
Description: Anti-HPV-16/18 antibody titers are presented as Geometric Mean Titers (GMTs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
  The immune response of the HPV-16/18 vaccine (as determined by anti-HPV-16/18 antibodies assessed by ELISA) in the HPV-060 study population was compared with the immune response obtained in study HPV-001 and its long-term follow-up studies HPV-007/HPV-023 at equivalent timepoints and with the immune response obtained after natural infection in subjects from study HPV-008.
  The immune response data for the efficacy studies HPV-001/HPV-007/HPV-023 can be found under the NCT record NCT00518336. The immune response data for the HPV-008 study can be found under the NCT record NCT00122681.
Time Frame: At Years 5, 6 and 7
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity at Years 5, 6 and 7, which included all evaluable subjects from the ATP cohort for immunogenicity of the primary study HPV-014 (NCT00196937), who were seronegative before vaccination and for whom immunogenicity data at Years 5, 6 and 7 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 134 | 146 | 146
EL.U/mL
  Anti-HPV-16 [Year 5]: number analyzed (Participants) | 128 | 127 | 118
  Anti-HPV-16 [Year 5] | 1495.7 [1249.2 to 1790.9] | 518.7 [423.2 to 635.6] | 282.4 [234.3 to 340.5]
  Anti-HPV-16 [Year 6]: number analyzed (Participants) | 128 | 130 | 116
  Anti-HPV-16 [Year 6] | 1344.6 [1130.2 to 1599.6] | 526.0 [434.7 to 636.4] | 277.7 [228.0 to 338.2]
  Anti-HPV-16 [Year 7]: number analyzed (Participants) | 125 | 119 | 111
  Anti-HPV-16 [Year 7] | 1014.0 [847.0 to 1214.0] | 369.5 [295.7 to 461.7] | 201.4 [163.6 to 247.9]
  Anti-HPV-18 [Year 5]: number analyzed (Participants) | 134 | 144 | 146
  Anti-HPV-18 [Year 5] | 440.4 [367.8 to 527.2] | 168.8 [140.7 to 202.4] | 104.6 [86.0 to 127.2]
  Anti-HPV-18 [Year 6]: number analyzed (Participants) | 133 | 146 | 142
  Anti-HPV-18 [Year 6] | 438.2 [366.6 to 523.7] | 167.5 [138.1 to 203.1] | 97.6 [79.2 to 120.3]
  Anti-HPV-18 [Year 7]: number analyzed (Participants) | 130 | 136 | 137
  Anti-HPV-18 [Year 7] | 307.8 [256.2 to 369.7] | 119.8 [98.4 to 145.9] | 81.7 [65.7 to 101.5]

2. Primary Outcome: Anti-HPV-16/18 Antibody Titers in Serum at Years 8, 9 and 10
Description: Anti-HPV-16/18 antibody titers are presented as Geometric Mean Titers (GMTs) and expressed in EL.U/mL.
  The immune response of the HPV-16/18 vaccine (as determined by anti-HPV-16/18 antibodies assessed by ELISA) in the HPV-060 study population was compared with the immune response obtained in study HPV-001 and its long-term follow-up studies HPV-007/HPV-023 at equivalent timepoints and with the immune response obtained after natural infection in subjects from study HPV-008.
  The immune response data for the efficacy studies HPV-001/HPV-007/HPV-023 can be found under the NCT number NCT00518336. The immune response data for the HPV-008 study can be found under the NCT number NCT00122681.
Time Frame: At Years 8, 9 and 10
Population: The analysis was performed on the ATP cohort for immunogenicity at Years 8, 9 and 10, which included all evaluable subjects from the ATP cohort for immunogenicity of the primary study HPV-014 (NCT00196937), who were seronegative before vaccination and for whom immunogenicity data at Years 8, 9 and 10 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 132 | 148 | 132
EL.U/mL
  Anti-HPV-16 [Year 8]: number analyzed (Participants) | 116 | 106 | 99
  Anti-HPV-16 [Year 8] | 1123.3 [930.2 to 1356.5] | 392.1 [315.3 to 487.7] | 189.1 [153.0 to 233.7]
  Anti-HPV-16 [Year 9]: number analyzed (Participants) | 127 | 132 | 110
  Anti-HPV-16 [Year 9] | 980.9 [825.5 to 1165.6] | 366.5 [303.5 to 442.6] | 180.2 [148.4 to 218.7]
  Anti-HPV-16 [Year 10]: number analyzed (Participants) | 123 | 121 | 107
  Anti-HPV-16 [Year 10] | 965.4 [802.2 to 1161.8] | 334.4 [270.5 to 413.5] | 157.4 [128.4 to 193.1]
  Anti-HPV-18 [Year 8]: number analyzed (Participants) | 120 | 123 | 120
  Anti-HPV-18 [Year 8] | 375.1 [310.6 to 453.0] | 134.1 [107.5 to 167.4] | 82.6 [65.9 to 103.6]
  Anti-HPV-18 [Year 9] | 327.4 [273.4 to 392.1] | 122.5 [101.1 to 148.4] | 75.6 [60.9 to 94.0]
  Anti-HPV-18 [Year 10]: number analyzed (Participants) | 127 | 142 | 130
  Anti-HPV-18 [Year 10] | 321.1 [265.0 to 389.1] | 115.4 [93.9 to 142.0] | 69.7 [56.0 to 86.8]

3. Primary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies at Years 5, 6 and 7
Description: Seroconversion was defined as the appearance of anti-HPV-16 and anti- HPV-18 antibodies [i.e. antibody titer greater than or equal to (≥) the cut-off value] in the serum of subjects seronegative before vaccination in the primary study HPV-014 (NCT00196937). Cut-off values were 8 EL.U/mL for anti-HPV-16 antibody titers and 7 EL.U/mL for anti-HPV-18 antibody titers.
Time Frame: At Years 5, 6 and 7
Population: The analysis was performed on the ATP cohort for immunogenicity at Years 5, 6 and 7, which included all evaluable subjects from the ATP cohort for immunogenicity of the primary study HPV-014 (NCT00196937), who were seronegative before vaccination and for whom immunogenicity data at Years 5, 6 and 7 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 134 | 146 | 146
Participants
  anti-HPV-16 [Year 5]: number analyzed (Participants) | 128 | 127 | 118
  anti-HPV-16 [Year 5] | 128 | 127 | 118
  anti-HPV-16 [Year 6]: number analyzed (Participants) | 128 | 130 | 116
  anti-HPV-16 [Year 6] | 128 | 130 | 116
  anti-HPV-16 [Year 7]: number analyzed (Participants) | 125 | 119 | 111
  anti-HPV-16 [Year 7] | 125 | 119 | 111
  anti-HPV-18 [Year 5]: number analyzed (Participants) | 134 | 144 | 146
  anti-HPV-18 [Year 5] | 134 | 144 | 143
  anti-HPV-18 [Year 6]: number analyzed (Participants) | 133 | 146 | 142
  anti-HPV-18 [Year 6] | 133 | 146 | 138
  anti-HPV-18 [Year 7]: number analyzed (Participants) | 130 | 136 | 137
  anti-HPV-18 [Year 7] | 130 | 135 | 131

4. Primary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies at Years 8, 9 and 10
Description: Seroconversion was defined as the appearance of anti-HPV-16 and anti-HPV-18 antibodies (i.e. antibody titer ≥ the cut-off value) in the serum of subjects seronegative before vaccination in the primary study HPV-014 (NCT00196937). Cut-off values were 19 EL.U/mL for anti-HPV-16 antibody titers and 18 EL.U/mL for anti-HPV-18 antibody titers.
Time Frame: At Years 8, 9 and 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 132 | 148 | 132
Participants
  anti-HPV-16 [Year 8]: number analyzed (Participants) | 116 | 106 | 99
  anti-HPV-16 [Year 8] | 116 | 106 | 95
  anti-HPV-16 [Year 9]: number analyzed (Participants) | 127 | 132 | 110
  anti-HPV-16 [Year 9] | 127 | 132 | 106
  anti-HPV-16 [Year 10]: number analyzed (Participants) | 123 | 121 | 107
  anti-HPV-16 [Year 10] | 123 | 120 | 103
  anti-HPV-18 [Year 8]: number analyzed (Participants) | 120 | 123 | 120
  anti-HPV-18 [Year 8] | 120 | 118 | 104
  anti-HPV-18 [Year 9] | 132 | 141 | 113
  anti-HPV-18 [Year 10]: number analyzed (Participants) | 127 | 142 | 130
  anti-HPV-18 [Year 10] | 126 | 133 | 109

5. Secondary Outcome: Anti-HPV-16/18 Secretion Antibody Titers in Cervico-vaginal Secretion (CVS) Samples at Years 5 and 6 in a Subset of Subjects
Description: Anti-HPV-16/18 titers in CVS samples are presented as GMTs and expressed in EL.U/mL.
Time Frame: At Year 5 and Year 6
Population: Analysis was performed on a subset of subjects from the Total Vaccinated Cohort (TVC), who volunteered for CVS sample collection at Years 5 and 6 and for whom the collected CVS sample contained less than 200 erythrocytes per microliter.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 39 | 39 | 28
EL.U/mL
  Anti-HPV-16 [Year 5] | 90.2 [61.9 to 131.3] | 47.2 [32.2 to 69.2] | 56.8 [28.7 to 112.4]
  Anti-HPV-18 [Year 5] | 30.9 [20.9 to 45.6] | 24.6 [14.8 to 41.0] | 33.3 [15.8 to 70.0]
  Anti-HPV-16 [Year 6]: number analyzed (Participants) | 29 | 29 | 26
  Anti-HPV-16 [Year 6] | 80.3 [46.8 to 137.8] | 43.8 [26.0 to 73.9] | 37.1 [20.8 to 66.0]
  Anti-HPV-18 [Year 6]: number analyzed (Participants) | 29 | 29 | 26
  Anti-HPV-18 [Year 6] | 22.9 [13.8 to 37.9] | 19.9 [11.4 to 34.9] | 19.2 [11.7 to 31.8]

6. Secondary Outcome: Anti-HPV-16/18 Secretion Antibody Titers in CVS Samples at Years 7, 8, 9 and 10 in a Subset of Subjects
Description: Anti-HPV-16/18 titers in CVS samples are presented as GMTs and expressed in EL.U/mL.
Time Frame: At Years 7, 8, 9 and 10
Population: Analysis was performed on a subset of subjects from the TVC, who volunteered for CVS sample collection at Years 7, 8, 9 and 10 and for whom the collected CVS sample contained less than 200 erythrocytes per microliter.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 41 | 40 | 32
EL.U/mL
  Anti-HPV-16 [Year 7]: number analyzed (Participants) | 31 | 30 | 30
  Anti-HPV-16 [Year 7] | 63.0 [38.6 to 102.9] | 33.3 [21.6 to 51.2] | 42.3 [25.0 to 71.5]
  Anti-HPV-18 [Year 7]: number analyzed (Participants) | 31 | 31 | 30
  Anti-HPV-18 [Year 7] | 33.5 [19.8 to 56.6] | 17.5 [10.2 to 30.1] | 49.0 [22.4 to 107.3]
  Anti-HPV-16 [Year 8]: number analyzed (Participants) | 31 | 34 | 32
  Anti-HPV-16 [Year 8] | 45.6 [29.6 to 70.1] | 43.9 [24.8 to 77.7] | 54.6 [34.3 to 86.8]
  Anti-HPV-18 [Year 8]: number analyzed (Participants) | 31 | 34 | 32
  Anti-HPV-18 [Year 8] | 17.8 [11.2 to 28.4] | 26.2 [14.7 to 46.8] | 31.9 [14.7 to 69.2]
  Anti-HPV-16 [Year 9]: number analyzed (Participants) | 32 | 35 | 27
  Anti-HPV-16 [Year 9] | 67.7 [45.4 to 101.0] | 42.6 [23.6 to 76.8] | 62.6 [36.7 to 106.5]
  Anti-HPV-18 [Year 9]: number analyzed (Participants) | 32 | 35 | 27
  Anti-HPV-18 [Year 9] | 28.1 [18.5 to 42.8] | 23.9 [15.8 to 36.1] | 50.4 [25.1 to 101.3]
  Anti-HPV-16 [Year 10]: number analyzed (Participants) | 41 | 40 | 26
  Anti-HPV-16 [Year 10] | 43.4 [28.1 to 67.1] | 34.3 [24.1 to 48.7] | 56.0 [31.5 to 99.7]
  Anti-HPV-18 [Year 10]: number analyzed (Participants) | 41 | 40 | 26
  Anti-HPV-18 [Year 10] | 29.4 [17.6 to 49.4] | 22.7 [13.8 to 37.3] | 45.1 [22.9 to 88.6]

7. Secondary Outcome: Total Immunoglobulin G (IgG) Secretion Antibody Titers in CVS Samples at Years 5 and 6 in a Subset of Subjects
Description: IgG antibody titers in CVS samples are presented as GMTs and expressed in microgram per milliliter (µg/mL).
Time Frame: At Year 5 and Year 6
Population: Analysis was performed on a subset of subjects from the TVC, who volunteered for CVS sample collection at Year 5 and Year 6 and for whom the collected CVS sample contained less than 200 erythrocytes per microliter.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 39 | 39 | 28
µg/mL
  IgG secretion antibodies [Year 5] | 577.8 [411.3 to 811.6] | 550.5 [373.7 to 811.0] | 990.6 [540.2 to 1816.4]
  IgG secretion antibodies [Year 6]: number analyzed (Participants) | 29 | 29 | 26
  IgG secretion antibodies [Year 6] | 546.5 [352.2 to 848.2] | 499.8 [327.7 to 762.2] | 1012.9 [696.7 to 1472.6]

8. Secondary Outcome: Total IgG Secretion Antibody Titers in CVS Samples at Years 7, 8, 9, and 10 in a Subset of Subjects
Description: Total IgG antibody titers in CVS samples are presented as GMTs and expressed in microgram per milliliter (µg/mL).
Time Frame: At Years 7, 8, 9 and 10
Population: Analysis was performed on a subset of subjects from the TVC, who volunteered for CVS sample collection at Years 7, 8, 9, 10 and for whom the collected CVS sample contained less than 200 erythrocytes per microliter.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 39 | 37 | 32
µg/mL
  IgG secretion antibodies [Year 7]: number analyzed (Participants) | 31 | 31 | 30
  IgG secretion antibodies [Year 7] | 517.5 [348.1 to 769.4] | 372.2 [236.7 to 585.4] | 1263.2 [793.8 to 2010.2]
  IgG secretion antibodies [Year 8]: number analyzed (Participants) | 31 | 34 | 32
  IgG secretion antibodies [Year 8] | 304.8 [211.1 to 440.1] | 457.2 [308.2 to 678.2] | 928.2 [578.0 to 1490.6]
  IgG secretion antibodies [Year 9]: number analyzed (Participants) | 32 | 33 | 26
  IgG secretion antibodies [Year 9] | 435.1 [293.2 to 645.8] | 460.4 [301.7 to 702.4] | 925.8 [586.3 to 1461.8]
  IgG secretion antibodies [Year 10]: number analyzed (Participants) | 39 | 37 | 24
  IgG secretion antibodies [Year 10] | 315.3 [237.9 to 417.8] | 373.5 [259.9 to 536.8] | 622.9 [405.2 to 957.5]

9. Secondary Outcome: Total IgG Antibody Titers in Serum at Years 5, 6 and 7 Based on the ATP Cohort for Immunogenicity
Description: Total IgG antibody titers are presented as GMTs and expressed in µg/mL.
Time Frame: At Years 5, 6 and 7
Population: The analysis was performed on the ATP cohort for immunogenicity at Years 5, 6 and 7, which included all evaluable subjects from the ATP cohort for immunogenicity of the primary study HPV-014 (NCT00196937) and for whom immunogenicity data at Years 5, 6 and 7 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 68 | 65 | 60
µg/mL
  Total IgG serum antibodies [Year 5] | 19481.8 [18076.2 to 20996.8] | 18388.2 [16844.6 to 20073.3] | 17657.2 [16046.7 to 19429.4]
  Total IgG serum antibodies [Year 6]: number analyzed (Participants) | 41 | 38 | 33
  Total IgG serum antibodies [Year 6] | 13376.5 [12498.7 to 14315.9] | 12262.7 [11304.8 to 13301.8] | 12040.2 [10854.4 to 13355.7]
  Total IgG serum antibodies [Year 7]: number analyzed (Participants) | 59 | 63 | 57
  Total IgG serum antibodies [Year 7] | 13957.2 [13116.6 to 14851.7] | 13179.4 [12287.7 to 14135.7] | 12992.9 [12096.9 to 13955.4]

10. Secondary Outcome: Total IgG Antibody Titers in Serum at Years 8, 9 and 10 Based on the ATP Cohort for Immunogenicity
Description: Total IgG antibody titers are presented as GMTs and expressed in µg/mL.
Time Frame: At Years 8, 9 and 10
Population: The analysis was performed on the ATP cohort for immunogenicity at Years 8, 9 and 10, which included all evaluable subjects from the ATP cohort for immunogenicity of the primary study HPV-014 (NCT00196937) and for whom immunogenicity data at Years 8, 9 and 10 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 61 | 62 | 55
µg/mL
  Total IgG serum antibodies [Year 8]: number analyzed (Participants) | 57 | 58 | 55
  Total IgG serum antibodies [Year 8] | 11059.5 [10547.8 to 11596.0] | 10656.3 [10057.6 to 11290.6] | 10605.7 [10061.4 to 11179.5]
  Total IgG serum antibodies [Year 9]: number analyzed (Participants) | 60 | 56 | 54
  Total IgG serum antibodies [Year 9] | 11212.2 [10661.3 to 11791.6] | 10693.8 [10067.0 to 11359.7] | 10427.8 [9871.3 to 11015.6]
  Total IgG serum antibodies [Year 10]: number analyzed (Participants) | 61 | 62 | 51
  Total IgG serum antibodies [Year 10] | 11071.3 [10546.9 to 11621.8] | 10650.8 [10079.2 to 11254.7] | 10535.0 [9979.4 to 11121.5]

11. Secondary Outcome: Total IgG Antibody Titers in Serum at Years 5, 6 and 7 Based on the TVC
Description: Total IgG antibody titers are presented as GMTs and expressed in µg/mL.
Time Frame: At Years 5, 6 and 7
Population: The analysis was performed on the TVC at Years 5, 6 and 7, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data at Years 5, 6 and 7 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 69 | 68 | 61
µg/mL
  Total IgG serum antibodies [Year 5] | 19453.0 [18068.5 to 20943.6] | 18092.4 [16566.3 to 19759.1] | 17885.0 [16224.1 to 19715.9]
  Total IgG serum antibodies [Year 6]: number analyzed (Participants) | 42 | 39 | 33
  Total IgG serum antibodies [Year 6] | 13318.5 [12458.3 to 14238.1] | 12173.1 [11231.2 to 13193.9] | 12040.2 [10854.4 to 13355.7]
  Total IgG serum antibodies [Year 7]: number analyzed (Participants) | 59 | 66 | 58
  Total IgG serum antibodies [Year 7] | 13957.2 [13116.6 to 14851.7] | 13059.5 [12205.2 to 13973.6] | 13052.9 [12160.9 to 14010.5]

12. Secondary Outcome: Total IgG Antibody Titers in Serum at Years 8, 9 and 10 Based on the TVC
Description: Total IgG antibody titers are presented as GMTs and expressed in µg/mL.
Time Frame: At Years 8, 9 and 10
Population: The analysis was performed on the Total Vaccinated Cohort at Years 8, 9 and 10, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data at Years 8, 9 and 10 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 62 | 66 | 57
µg/mL
  Total IgG serum antibodies [Year 8]: number analyzed (Participants) | 58 | 61 | 57
  Total IgG serum antibodies [Year 8] | 11084.4 [10578.2 to 11614.8] | 10602.4 [10010.8 to 11229.1] | 10725.5 [10151.1 to 11332.4]
  Total IgG serum antibodies [Year 9]: number analyzed (Participants) | 60 | 56 | 54
  Total IgG serum antibodies [Year 9] | 11212.2 [10661.3 to 11791.6] | 10693.8 [10067.0 to 11359.7] | 10427.8 [9871.3 to 11015.6]
  Total IgG serum antibodies [Year 10]: number analyzed (Participants) | 62 | 66 | 55
  Total IgG serum antibodies [Year 10] | 11043.6 [10526.3 to 11586.4] | 10511.3 [9938.6 to 11117.0] | 10484.8 [9947.5 to 11051.1]

13. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 4 in Primary Study HPV-014 (NCT00196937) to Year 5 in the Present Study
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject, or may have evolved into one of the outcomes listed above. Related SAE = SAE assessed by the investigator as causally related to the study vaccine administered in study HPV-014 (NCT00196937).
Time Frame: From Year 4 in primary study HPV-014 (NCT00196937) up to Year 5 in present HPV-060 study
Population: The analysis was based on the TVC at Year 5, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 153 | 184 | 170
Participants
  Fatal SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 5 to Year 6
Description: as for outcome 13
Time Frame: From Year 5 up to Year 6
Population: The analysis was based on the TVC at Year 6, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 147 | 177 | 164
Participants
  Fatal SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 6 to Year 7
Description: as for outcome 13
Time Frame: From Year 6 up to Year 7
Population: The analysis was based on the TVC at Year 7, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 149 | 165 | 160
Participants
  Fatal SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 7 to Year 8
Description: as for outcome 13
Time Frame: From Year 7 up to Year 8
Population: The analysis was based on the TVC at Year 8, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 137 | 152 | 141
Participants
  Fatal SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 8 to Year 9
Description: as for outcome 13
Time Frame: From Year 8 up to Year 9
Population: The analysis was based on the TVC at Year 9, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 9.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 146 | 180 | 157
Participants
  Fatal SAE(s) | 0 | 0 | 1
  Related SAE(s) | 0 | 1 | 0

18. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 9 to Year 10
Description: as for outcome 13
Time Frame: From Year 9 up to Year 10
Population: The analysis was based on the TVC at Year 10, which included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available at Year 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 142 | 172 | 156
Participants
  Fatal SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 1 | 0

19. Secondary Outcome: Number of Subjects With Any Fatal or Vaccine-related SAEs (Including SAEs Related to Study Procedures and GlaxoSmithKline Biologicals' Concomitant Medication) From Year 0 to Year 10
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject. Related SAE = SAE assessed by the investigator as causally related to the study vaccine administered in study HPV-014 (NCT00196937).
Time Frame: From Year 0 up to Year 10
Population: The analysis was performed on the TVC that included all vaccinated subjects [i.e. all subjects who received 3 doses of HPV vaccine in the primary study HPV-014 (NCT00196937)] for whom data were available throughout the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
Number analyzed (Participants) | 159 | 194 | 171
Participants
  Fatal SAE(s) | 0 | 1 | 1
  Related SAE(s) | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs: Throughout the entire study period (from Year 0 up to the Year 10).
Description: Other (non-serious) Adverse Events and solicited symptoms were not collected/assessed. This section displays the safety analysis on the subjects who participated in the primary study HPV-014 (NCT00196937), excluding those who were not selected or not consented for the present study HPV-060 (NCT00947115).
Arm/Group | Cervarix 15-25 Years Group | Cervarix 26-45 Years Group | Cervarix 46-55 Years Group
All-Cause Mortality (participants affected / at risk) | 0/159 | 1/194 | 1/171
Serious Adverse Events (participants affected / at risk) | 0/159 | 2/194 | 1/171
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix 15-25 Years Group (N=159) | Cervarix 26-45 Years Group (N=194) | Cervarix 46-55 Years Group (N=171)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cervical displasia (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.